CLINICAL TRIAL: NCT00694993
Title: A Double-blind, Placebo-controlled, Randomized Single Dose Escalation Study and a Double-blind, Placebo-controlled, Randomised Parallel Group 14-days Once Daily Repeat Dose Study to Investigate Safety, Tolerability and Pharmacokinetics of an Intranasal H1/H3 Dual Antagonist Compound in Healthy Male Subjects
Brief Title: Single and Repeat Dose First Time in Human Study for an Intranasal H1/H3 Dual Antagonist in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Purpose: Treatment
Other Study IDs: HHI110157
Record Dates: First submitted 2008-06-09; First posted 2008-06-11 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Rhinitis, Allergic, Seasonal
Keywords: first time in human; Allergic rhinitis,
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis, Allergic | interventions — GSK 1004723

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Subjects receiving GSK1004723 + placebo in cohort I and II (Experimental): Eligible subjects will receive GSK1004723 nasal spray with single doses of 50 micrograms, 100 micrograms, 200 micrograms, 500 micrograms and 1000 micrograms. Subjects will also receive placebo nasal spray.
  Interventions: Drug: GSK1004723; Drug: Placebo
- Subjects receiving GSK1004723 200 micrograms in cohort III (Experimental): Eligible subjects will receive nasal spray of GSK1004723 with escalated repeat doses of 200 micrograms given once daily for 14 days.
  Interventions: Drug: GSK1004723
- Subjects receiving placebo in cohort III (Experimental): Eligible subjects will receive nasal spray of placebo given once daily for 14 days.
  Interventions: Drug: Placebo
- Subjects receiving GSK1004723 1000 micrograms in cohort IV (Experimental): Eligible subjects will receive nasal spray of GSK1004723 with escalated repeat doses of 1000 micrograms given once daily for 14 days.
  Interventions: Drug: GSK1004723
- Subjects receiving placebo in cohort IV (Experimental): Eligible subjects will receive nasal spray of placebo given once daily for 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK1004723 — GSK1004723 will be supplied as intranasal sprays aqueous suspensions for intranasal spray administration.
  Arms: Subjects receiving GSK1004723 + placebo in cohort I and II; Subjects receiving GSK1004723 1000 micrograms in cohort IV; Subjects receiving GSK1004723 200 micrograms in cohort III
Drug: Placebo — Placebo will be supplied as intranasal sprays aqueous suspensions for intranasal spray administration.
  Arms: Subjects receiving GSK1004723 + placebo in cohort I and II; Subjects receiving placebo in cohort III; Subjects receiving placebo in cohort IV

SUMMARY:
This is a double-blind, placebo-controlled, randomized single dose escalation study and a double-blind, placebo-controlled, randomised parallel group 14-days once daily repeat dose study to investigate safety, tolerability and pharmacokinetics of an intranasal H1/H3 dual antagonist compound in healthy male subjects.

DETAILED DESCRIPTION:
A double-blind, placebo-controlled, randomized single dose escalation study and a double-blind, placebo-controlled, randomised parallel group 14-days once daily repeat dose study to investigate safety, tolerability and pharmacokinetics of an intranasal H1/H3 dual antagonist compound in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects aged between 18 and 50 years inclusive.
* Body mass index within the range 19-29.9kg/m2 (inclusive), with weight range of 50 kg-100 kg (inclusive).
* Healthy (defined as individuals who are free from significant nasal, cardiac, pulmonary, gastrointestinal, hepatic, renal, haematological, malignancy, endocrine, neurological and psychiatric disease as determined by history, physical examination and screening investigations).
* Non-smoking status as verified by urinary cotinine levels below 500 ng/mL cotinine at the screening visit. This can include ex-smokers who have given up smoking for >1 year.
* Normal nasal examination as per Ear, Nose and Throat (ENT) assessment
* No significant ECG abnormalities and QTc (B) <450 msec.
* The subject is able and willing to give written informed consent to take part in the study and is available to complete all study measurements.
* Male subjects must agree to abstain from or use a condom during sexual intercourse with female partners of childbearing potential, to prevent either pregnancy in the female partner or the possible exposure of a pregnant or lactating female to the investigational product from the male subject's semen. In addition, female partners of male subjects must use a reliable contraceptive method listed in the protocol, or they must refrain from sexual intercourse from the first dose of study medication until 84 days after the last dose.

Exclusion Criteria:

* As a result of the medical interview, physical examination or screening investigations, the Investigator or appropriately qualified designee considers the subject unfit for the study.
* The subject has a history of drug or any other allergy, which, in the opinion of the Investigator or appropriately qualified designee, contraindicates their participation, including known or suspected personal history or family history of adverse reactions or hypersensitivity to anti histamines
* The subject has participated in a study with a new molecular entity during the previous 3 months or any other study during the previous 2 months.
* The subject regularly, or on average, drinks more than 21 units of alcohol a week or more than an average intake of 3 units per day.
* The subject is currently taking regular (or a course of) medication, prescribed (including all beta-agonists) or not (including over the counter medication or herbal remedies such as St Johns Wort). Paracetamol is an exception and will be permitted at daily doses of up to 4g following the first dose of investigational product.
* The subject has tested positive for hepatitis C antibody or hepatitis B surface antigen.
* The subject has tested positive for HIV.
* The subject has a positive drugs of abuse and alcohol test.
* Donation during the study would result in >500mL of blood being donated over a 56 day period
* Subjects with structural nasal abnormalities frequent nose bleeds, Perennial Allergic Rhinitis (PAR) and Seasonal Allergic Rhinitis (SAR) unless subjects with SAR are asymptomatic and it is outside of the pollen season
* Subjects who are unable to comply with study procedures
* Subject is the Investigator or any sub-investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the study
* Vulnerable subjects (eg. persons kept in detention)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2007-12-17 (Actual); Primary Completion 2008-05-26 (Actual); Study Completion 2008-05-26 (Actual)

PRIMARY OUTCOMES:
ECG monitoring during 24 hours after each dose in the single dose cohorts and on days 1 and 7 in the repeat dose cohorts. | during 24 hours after each dose in the single dose cohorts and on days 1 and 7 in the repeat dose cohorts
Heart rate and blood pressure changes over 24 hours after dosing in single and repeat dose cohorts | over 24 hours after dosing

SECONDARY OUTCOMES:
Blood drug levels for GSK1004723 following single and repeat intranasal dosing | Pre-dose, 15 minutes, 30 minutes, 45 minutes, 1 hour, 2 hours, 4 hours, 6 hours, 8 hours, 12 hours and 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Daley-Yates P, Ambery C, Sweeney L, Watson J, Oliver A, McQuade B. The efficacy and tolerability of two novel H(1)/H(3) receptor antagonists in seasonal allergic rhinitis. Int Arch Allergy Immunol. 2012;158(1):84-98. doi: 10.1159/000329738. Epub 2011 Dec 29. PMID 22212854
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study HHI110157 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/HHI110157?search=study&study_ids=HHI110157#rs
- Available data/document: Study Protocol: HHI110157 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: HHI110157 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: HHI110157 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: HHI110157 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: HHI110157 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: HHI110157 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: HHI110157 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register